CLINICAL TRIAL: NCT06610500
Title: Clozapine Hematological Monitoring Regulatory Compliance Assessment in Psychiatry
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN682023/CHUSTE
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Schizophrenia; Agranulocytosis
Keywords: Clozapine; schizophrenia; hematological monitoring; agranulocytosis; regulation; paper tracking book
MeSH Terms: conditions — Schizophrenia; Agranulocytosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Population 1: Patients treated and stabilised by clozapine in the active queue of Medical-Psychological Center (CMP) of St-Etienne
  Interventions: Other: Questionnaires
- Population 2: Liberal psychiatrists practising in the Loire department, and hospital psychiatrists
  Interventions: Other: Questionnaires
- Population 3: Pharmacists practising in community pharmacies dispensing clozapine to patients, hospital Pharmacists in the Loire
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires investigating the prescription and dispensing of clozapine.

SUMMARY:
Clozapine is a drug that requires regular and diligent hematological monitoring throughout its use. This follow-up is, in France, framed by a compulsory paper format of the blood count follow-up notebook for each patient. Due to the multiplicity of the different modes of transmission of the different documents necessary for compliance with the regulations for the prescription, dispensing and administration of clozapine, we decided to carry out a current inventory in the department of Loire with respect for the latter. The main objective of this study is to assess the rate of non-compliance in circuits of prescription, dispensing and administration of clozapine by sending a questionnaire on habits of prescriptions, dispensing and administration of health professionals (psychiatrists, pharmacists), and by sending a questionnaire to the patients treated by clozapine.

ELIGIBILITY:
Inclusion Criteria:

* Population 1: all patients stabilized of Medical-Psychological Center (CMP) of St-Etienne treated with clozapine
* Population 2 : all psychiatrists of the Loire department
* Population 2 : all pharmacists of the Loire department

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated and stabilised on clozapine by the St-Etienne Psychiatry Department Private and hospital psychiatrists in the Loire Pharmacists and hospital pharmacists in the Loire
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Rate of non-compliance | Month: 2
  Rate of non-compliance in the circuits for prescribing, dispensing clozapine

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Cécile GALLO BLANDIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No